CLINICAL TRIAL: NCT05405920
Title: Implementing and Scaling Up a Team-based Care Strategy for Hypertension Control in Colombia and Jamaica
Brief Title: Caribbean and South America Team-based Strategy to Control Hypertension
Acronym: CATCH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Universidad de Santander (Other); University of the West Indies, Jamaica (Unknown)
Responsible Party: Principal Investigator, Jiang He, MD, PhD, Professor and Chair, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UG3HL152373 (NIH)
Record Dates: First submitted 2022-05-27; First posted 2022-06-06 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: cluster-randomization of 40 primary care clinics
Masking Description: Due to the nature of the cluster design and intervention program, the study participants, primary care physicians, nurses, community health workers, and research staff who collected clinical outcome data will not be blinded. The outcome adjudication committee members, however, will be blinded to randomization assignment for adverse event evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Team-based Care Strategy for Hypertension Control (Experimental): The core component of the intervention is a stepped-care protocol, based on the 2017 American College of Cardiology (ACC)/American Heart Association (AHA) Clinical Practice Guideline for High Blood Pressure and the 2021 World Health Organization (WHO) Hypertension Guideline. Using a team-based care model, a physician-nurse-CHW team will work with patients to implement clinical guideline-based treatment in all intervention clinics. Team-based care components will include task sharing and shifting, health care team training, home BP monitoring, BP audit and feedback, and CHW-led health coaching on lifestyle modification and medication adherence.
  Interventions: Behavioral: Team-based Care Strategy for Hypertension Control
- Enhanced Usual Care (Active Comparator): We will train the primary care physicians, nurses, and other clinic staff in performing standardized BP measurements. We will offer physician education on clinical guidelines for hypertension management and issue continuing medical education credits. Patient educational materials will be distributed. We will not conduct any other interventions in the enhanced usual care clinics.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Team-based Care Strategy for Hypertension Control — The core component of the intervention is a stepped-care protocol, based on the 2017 American College of Cardiology (ACC)/American Heart Association (AHA) Clinical Practice Guideline for High Blood Pressure and the 2021 World Health Organization (WHO) Hypertension Guideline. Using a team-based care model, a physician-nurse-CHW team will work with patients to implement clinical guideline-based treatment in all intervention clinics. Team-based care components will include task sharing and shifting, health care team training, home BP monitoring, BP audit and feedback, and CHW-led health coaching on lifestyle modification and medication adherence.
  Arms: Team-based Care Strategy for Hypertension Control
Behavioral: Enhanced Usual Care — We will train the primary care physicians, nurses, and other clinic staff in performing standardized BP measurements. We will offer physician education on clinical guidelines for hypertension management and issue continuing medical education credits. Patient educational materials will be distributed. We will not conduct any other interventions in the enhanced usual care clinics.
  Arms: Enhanced Usual Care

SUMMARY:
The CATCH cluster randomized trial will test the implementation and effectiveness outcomes of implementing and scaling up a team-based care strategy for blood pressure control in Colombia and Jamaica.

DETAILED DESCRIPTION:
The CATCH Study includes a two-year UG3 Planning Phase and a four-year UH3 Implementation Phase. In the UH3 Implementation Phase, we will first conduct a cluster randomized implementation trial to test the effectiveness and implementation of a team-based care strategy for hypertension control among patients with hypertension in 40 clinics from Colombia and Jamaica (20 in each country). Twenty clinics will be randomized to the team-based care intervention and 20 to provider training intervention. A total of 1,680 patients (42 per clinic) with uncontrolled hypertension will be recruited into the study and followed for 18 months for effectiveness and implementation outcomes. A post-intervention study visit will take place 6 months after the end of the 18-month intervention to evaluate the sustainability of the implementation strategies. We will subsequently conduct a pre- and post- scale-up comparison study to implement the team-based care strategy in all remaining public primary care clinics that provide chronic disease management in Jamaica and primary care clinics in the seven participating departments in Colombia. A pre- and post- scale-up comparison design will be used to assess barriers and implementation outcomes before and 12 months after the scale-up intervention at the clinic, primary care physician, nurse/pharmacist, and community health worker (CHW) levels.

ELIGIBILITY:
Inclusion criteria for clinics:

* Serving >300 hypertensive patients during the previous year
* Clinic visits and BP medications are free of charge to patients
* Not sharing physicians, nurses, pharmacists, or community health workers (CHWs) with other clinics

Inclusion criteria for participants:

* Men or women aged ≥ 21 years who receive primary care from participating clinics
* Average untreated BP ≥140/90 mm Hg among individuals without a history of clinical cardiovascular disease (CVD), chronic kidney disease (CKD), or diabetes; average untreated BP ≥130/80 mm Hg among individuals aged ≥65 years or those with clinical CVD, CKD, or diabetes; or average treated BP ≥130/80 mm Hg from six BP readings at two screening visits
* Not pregnant or planning to become pregnant in the next 18 months
* Able and willing to give informed consent
* No plans to change primary care clinic in the next 18 months
* Not an immediate family member of staff at the primary care clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Net difference in mean change of systolic blood pressure | 18 months
  Differences in mean change of systolic BP from baseline to 18 months between intervention and control groups

SECONDARY OUTCOMES:
Difference in blood pressure control (<130/80 mm Hg) | 18 months
  Difference in the proportion of patients with systolic BP <130 mm Hg and diastolic BP <80 mm Hg between intervention and control groups at 18 months
Net difference in mean change of diastolic blood pressure | 18 months
  Differences in mean change of diastolic BP from baseline to 18 months between intervention and control groups
Side effects | 18 months
  Differences in medication side effects between intervention and control groups will be assessed by survey. A list of common side effects associated with high blood pressure will be asked of participants to collect presence and frequency of side effects.
Health-related quality of life | 18 months
  Differences in health-related quality of life (measured by EQ-SD and SF-12) between intervention and control groups
Cost-effectiveness | 18 months
  Incremental direct costs per additional percentage of hypertension control

OTHER OUTCOMES:
Acceptability | 18 months
  Measured by validated survey
Adoption | Baseline
  Defined as % of clinics adopting intervention components
Appropriateness | 18 months
  Measured by validated survey
Feasibility (suitability) | Baseline
  Measured by validated survey
Fidelity | 18 months
  % of each intervention component delivered per protocol
Implementation Costs | 18 months
  Defined as all costs associated with implementation and assessed from administrative data
Penetrance | 18 months
  Defined as % of providers using the intervention approach
Sustainability | 18 months
  % of clinics maintaining intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He, MD, PhD, Principal Investigator — Tulane University; Marshall Tulloch-Reid, MBBS, DSc, Principal Investigator — University of the West Indies, Jamaica; Patricio López-Jaramillo, MD, PhD, Principal Investigator — Universidad de Santander
Locations (2):
- 20 primary care clinics in Colombia, Santander, Colombia
- 20 primary care clinics in Jamaica, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Yes
Our study data sharing plan will comply with all NIH policies for data sharing. Data sharing will be executed through the centralized NIH data repository and will be implemented in a timely manner. Study data, including data from baseline and follow-up visits, will be prepared for transmission to the NHLBI data repository - the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC). Data will be prepared by the study data manager/biostatistician and sent to the Program Official for review prior to release. These data will be free of identifiers that allow identification of individual research participants either directly or through "deductive disclosure." We are very open to sharing data enthusiastically with the general scientific community, since we also believe in the added value of other investigators working on these data.
Supporting Information: Study Protocol, SAP
Time Frame: Data sets will be submitted to the study's NHLBI Program Official no later than 3 years after the end of the final patient follow-up visit or 2 years after the main paper of the trial has been published, whichever comes first.
Access Criteria: We will offer, through our public access website, opportunities for outside investigators to collaborate with us using complete study data.
URL: https://www.catch-study.org/

REFERENCES:
- [Derived] Mills KT, Ferguson T, Lopez-Lopez JP, Duncan J, Lanza P, Marshall A, Reyes M, Chen J, Anderson AH, Whelton PK, Bailey A, Lindsay C, Sanchez G, Lopez-Jaramillo P, Tulloch-Reid M, He J. Caribbean and South American team-based strategy to control hypertension (CATCH): Rationale and study design of a cluster randomized trial. Am Heart J. 2025 Dec 17;294:107329. doi: 10.1016/j.ahj.2025.107329. Online ahead of print. PMID 41419163
- See also: CATCH Study Website — https://www.catch-study.org/